CLINICAL TRIAL: NCT03137082
Title: Guanfacine to Reduce Relapse Risk in Women With Alcohol Use Disorder (AUD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Helen Fox, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AA024880 (NIH)
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Abstinence
Keywords: Alcohol Use Disorder; Guanfacine; Stress; Craving; Gender; Relapse
MeSH Terms: conditions — Alcohol Abstinence; Alcoholism; Coitus; Recurrence | interventions — Guanfacine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guanfacine XR 3mgs/daily (Experimental): * Guanfacine XR tablet by mouth every 24 hours for 12 weeks
  * 21 day titration: 1 mg/d (day 1-7); 2mgs/d (day 7-21)
  * Full dose: 3mgs/d (day 21- day 70)
  * 2 week taper: 2mgs/d (day 71-77); 1mg/d (day 77-83)
  Interventions: Drug: Guanfacine XR 3mgs/daily
- Placebo (for guanfacine) (Placebo Comparator): * Guanfacine XR tablet by mouth every 24 hours for 12 weeks
  * 21 day titration: 1 mg/d (day 1-7); 2mgs/d (day 7-21)
  * Full dose: 3mgs/d (day 21- day 70)
  * 2 week taper: 2mgs/d (day 71-77); 1mg/d (day 77-83)
  Interventions: Drug: Placebo (for guanfacine)

INTERVENTIONS:
Drug: Guanfacine XR 3mgs/daily — Guanfacine 3mg tablet
  Other Names: Intuniv
  Arms: Guanfacine XR 3mgs/daily
Drug: Placebo (for guanfacine) — Sugar pill manufactured to mimic guanfacine tablets
  Other Names: Sugar pill
  Arms: Placebo (for guanfacine)

SUMMARY:
Guanfacine may preferentially reduce craving and improve cognitive control in women with Alcohol Use Disorder (AUD), compared to men. As these behaviors are related to relapse, the objectives of this study are to conduct a 10-week out-patient clinical trial to examine the effects of Guanfacine Extended Release (XR; 3mgs) versus placebo on drinking measures in women with AUD.

DETAILED DESCRIPTION:
Gender-specific variation in sympathetic sensitivity (Fox et al., 2014; Fox and Sinha, 2009; Cahill, 2003; Heinsbroek et al., 1991) may mean that guanfacine is particularly efficacious in attenuating drinking in women, rather than men with Alcohol Use Disorder (AUD). Thus, the investigators propose a double blind, placebo-controlled, 10-week randomized clinical trial to examine the effects of Guanfacine XR (3mgs/daily) versus placebo in 60 women with AUD. This will include twice weekly appointments comprising medical management and contingency management protocols, collection of urine, breathalyzer screens, and vitals. Measures of craving and mood will also be assessed. Parallel laboratory challenge studies will also be conducted both on admission to out-patient treatment and again following 4 weeks of treatment, in order to better elucidate the potentially therapeutic mechanisms of guanfacine. Participants will be exposed to a personal stress versus relaxing imagery condition, 1 condition per day, in a randomized order. Craving, anxiety, mood, cognitive control, heart rate and blood pressure (HRBP), and biological stress system markers will be assessed at baseline, following imagery and at various recovery timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Must meet Diagnostic and Statistical Manual of Mental Disorders-V (DSM- V) criteria for moderate to severe Alcohol Use Disorder (AUD),
* Must produce positive urine toxicology screens on admission to study
* Must demonstrate good health as verified by screening examination
* Must be able to read English and complete study evaluations
* Must be able to provide informed written and verbal consent

Exclusion Criteria:

* Meeting current use disorder for any other psychoactive substance, excluding nicotine.
* Having any other current Axis I psychiatric disorders or medical conditions requiring treatment or medication
* EKG evidence at baseline screening of any clinically significant conduction abnormalities including a Bazlett's QTc (corrected QT interval) of >470 msec.
* Must not be on monophasic contraceptives, nursing or pregnant.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Fox, PhD, Principal Investigator — Stony Brook University
Locations (1):
- The Health Sciences Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox HC, Morgan PT, Sinha R. Sex differences in guanfacine effects on drug craving and stress arousal in cocaine-dependent individuals. Neuropsychopharmacology. 2014 May;39(6):1527-37. doi: 10.1038/npp.2014.1. Epub 2014 Jan 7. PMID 24395021
- [Background] Fox HC, Sinha R. Sex differences in drug-related stress-system changes: implications for treatment in substance-abusing women. Harv Rev Psychiatry. 2009;17(2):103-19. doi: 10.1080/10673220902899680. PMID 19373619
- [Background] Heinsbroek RP, van Haaren F, Feenstra MG, Boon P, van de Poll NE. Controllable and uncontrollable footshock and monoaminergic activity in the frontal cortex of male and female rats. Brain Res. 1991 Jun 14;551(1-2):247-55. doi: 10.1016/0006-8993(91)90939-s. PMID 1913155
- [Background] Cahill L. Sex-related influences on the neurobiology of emotionally influenced memory. Ann N Y Acad Sci. 2003 Apr;985:163-73. doi: 10.1111/j.1749-6632.2003.tb07080.x. PMID 12724157
- [Derived] Konjusha A, Colzato L, Ghin F, Stock AK, Beste C. Auricular transcutaneous vagus nerve stimulation for alcohol use disorder: A chance to improve treatment? Addict Biol. 2022 Sep;27(5):e13202. doi: 10.1111/adb.13202. PMID 36001426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from flyers posted in and around Stony Brook Hospital and its outpatient facilities, in addition to advertisements on social media. The first participant was enrolled in July 2017 and the last in March 2020
Pre-assignment Details: Following consent, participants were scheduled for an eligibility intake (including clinical and physical assessments). If eligible, they were scheduled for a second intake which included completing baseline assessments of alcohol and substance use in addition to alcohol craving, mood, anxiety and emotion regulation. Of the 32 women consented, N=17 did not meet criteria and N=15 were eligible and randomized onto study medication.
Groups:
- Guanfacine XR 3mgs/Daily: * Guanfacine XR tablet by mouth every 24 hours for 12 weeks
  * 21 day titration: 1 mg/d (day 1-7); 2mgs/d (day 7-21)
  * Full dose: 3mgs/d (day 21- day 70)
  * 2 week taper: 2mgs/d (day 71-77); 1mg/d (day 77-83)
  Guanfacine XR 3mgs/daily: Guanfacine 3mg tablet
- Placebo (for Guanfacine): * Guanfacine XR tablet by mouth every 24 hours for 12 weeks
  * 21 day titration: 1 mg/d (day 1-7); 2mgs/d (day 7-21)
  * Full dose: 3mgs/d (day 21- day 70)
  * 2 week taper: 2mgs/d (day 71-77); 1mg/d (day 77-83)
  Placebo (for guanfacine): Sugar pill manufactured to mimic guanfacine tablets
Period: Overall Study
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Started | 8 | 7
Completed | 6 | 6
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 32 women were enrolled in the study. N=17 were not eligible, N=15 were randomized to study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.9 (15.8) | 48.3 (11.1) | 42.6 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 5 | 7 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 0
% no. of drinking days in last 3 months [Mean (Standard Deviation); unit: percentage of days] | 50.1 (36.0) | 66.5 (39.1) | 58.3 (37.6)
no. of drinks consumed per occasion [Mean (Standard Deviation); unit: drinks per occasion] | 4.75 (1.9) | 4.9 (4.2) | 4.8 (2.0)
% no. of binge drinking days in last 3 months [Mean (Standard Deviation); unit: % no. of binge drinking days] | 41.1 (28.7) | 35.4 (36.1) | 38.3 (32.4)
Depressive Symptomatology [Mean (Standard Deviation); unit: units on a scale] — Depressive symptomatology was measured using the Beck Depression Inventory (BDI). Possible scores range from 0 to 63, with scores of > 40 reflecting "extreme depression". Baseline scores were collected at one time-point.
  units on a scale | 17.6 (12.9) | 11.83 (9.0) | 14.7 (11.0)
no. of smokers (tobacco) [Number; unit: participants] | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days Abstinent
Description: Percentage of days abstinent across the 12-week trial was calculated using the Timeline follow Back.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
percentage of days abstinent | 74.7 (27.4) | 50.6 (26.5)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p < 0.03, Mixed Models Analysis

2. Primary Outcome: Percentage of Heavy Drinking Days
Description: Percentage of heavy drinking days across the 12-week trial was calculated using the Timeline follow Back.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage heavy drinking days
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
percentage heavy drinking days | 15.5 (26.7) | 30.6 (26.7)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.1, Mixed Models Analysis

3. Primary Outcome: Alcohol Consumption (Percentage of Negative Urines)
Description: Urine screening will be conducted twice per week across the trial.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of negative urines
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
percentage of negative urines | 45.3 (35.7) | 35.2 (19.4)

4. Secondary Outcome: Mood (Anxiety)
Description: The Anxiety subscale of the Profile of Mood States (POMS) was administered to assess anxiety. The subscale comprises 9 adjectives that describe anxiety-related feelings, and participants are required to rate the extent to which they are experiencing each feeling at that moment, from 0= not at all; 1= a little; 2= moderately; 3= quite a bit; 4= extremely. Possible scores range from 0 to 36, with higher scores representing higher levels of anxiety. Anxiety ratings were collected two times per week across twelve weeks (24 time-points). Each time-point represented change from baseline anxiety. The calculation here represents mean change from baseline values across the 12 weeks, where minus scores represent lower mean anxiety compared with baseline.
Time Frame: 2 times per week for 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -8.2 (8.2) | -0.75 (4.7)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.01, Mixed Models Analysis

5. Secondary Outcome: Mood (Depression)
Description: The Depression subscale of the Profile of Mood States (POMS) was administered to assess depression. The subscale comprises 15 adjectives that describe depression-related feelings, and participants are required to rate the extent to which they are experiencing each feeling at that moment, from 0= not at all; 1= a little; 2= moderately; 3= quite a bit; 4= extremely. Possible scores range from 0 to 60, with higher scores representing higher levels of depression. Depression ratings were collected two times per week across twelve weeks (24 time-points). Each time-point represented change from baseline depression. The calculation here represents mean change from baseline values across the 12 weeks, where minus scores represent lower mean depression compared with baseline.
Time Frame: 2 times per week for 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -13.9 (13.3) | 0.03 (5.2)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.001, Mixed Models Analysis

6. Secondary Outcome: Alcohol Craving
Description: The desire for using alcohol was assessed using a 10-point visual analog scale (VAS) in which 1 = 'not at all' and 10 = 'extremely high'. Alcohol craving ratings were collected two times per week across twelve weeks (24 time-points). Each time-point represented change from baseline alcohol craving. The calculation here represents mean change from baseline values across the 12 weeks, where minus scores represent lower mean alcohol craving compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -1.6 (1.4) | -1.9 (3.4)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.5, Mixed Models Analysis

7. Secondary Outcome: Emotion Regulation (Difficulties in Impulse Control)
Description: We used the Impulse Control Difficulties subscale (IMPULSE) of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in impulse control across the trial. The DERS was administered two times per week, and the IMPULSE subscale comprised 6 items with a potential score range of 6 to 30 with higher scores representing greater difficulties in impulse control. Each time-point represents change from baseline impulse control difficulties. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties in impulse control compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -2.8 (2.4) | 0.85 (3.2)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p < .03, Mixed Models Analysis

8. Secondary Outcome: Emotion Regulation (Difficulties With Engaging in Goal Related Behavior)
Description: We used the Difficulties in Engaging in Goal-Directed Behavior (GOALS) subscale of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in goal-directed behavior across the trial. The DERS was administered two times per week (24 time-points) and the GOALS subscale comprised 5 items with a potential score range of 5 to 25 with higher scores representing greater difficulties in engaging in goal-directed behavior. Each time-point represented change from baseline GOALS. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties in engaging in goal-directed behavior compared with baseline.
Time Frame: 12-week
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -3.0 (3.6) | 0.95 (2.2)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.1, Mixed Models Analysis

9. Secondary Outcome: Emotion Regulation (Difficulties With Emotional Clarity)
Description: We used the Lack of Emotional Clarity subscale (CLARITY) of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in emotional clarity across the trial. The DERS was administered two times per week, and the CLARITY subscale comprised 5 items with a potential score range of 5 to 25 with higher scores representing greater difficulties in emotional clarity. Each time-point represents change from baseline difficulties in emotional clarity. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties in emotional clarity compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
units on a scale | -2.3 (2.8) | -0.71 (2.3)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p < 0.3, Mixed Models Analysis

10. Secondary Outcome: Emotion Regulation (Limited Access to Emotion Regulation Strategies)
Description: We used the Limited Access to Emotion Regulation Strategies subscale (STRATEGIES) of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in ability to access emotion regulation strategies across the trial. The DERS was administered two times per week, and the STRATEGIES subscale comprised 8 items with a potential score range of 8 to 40 with higher scores representing greater difficulties in accessing emotion regulation strategies. Each time-point represents change from baseline STRATEGIES. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties in accessing emotion regulation strategies compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -5.1 (5.4) | -0.28 (5.4)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.04, Mixed Models Analysis

11. Secondary Outcome: Emotion Regulation (Difficulties With Emotional Awareness)
Description: We used the Lack of Emotional Awareness subscale (AWARENESS) of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in emotional awareness across the trial. The DERS was administered two times per week, and the AWARENESS subscale comprised of 6 items with a potential score range of 6 to 30 with higher scores representing greater a greater lack of emotional awareness. Each time-point represents change from baseline emotional awareness. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties in emotional awareness compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -1.6 (4.3) | -2.9 (5.1)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.4, Mixed Models Analysis

12. Secondary Outcome: Emotion Regulation (Non-Acceptance of Emotional Responses)
Description: We used the Non-Acceptance of Emotional Responses subscale (NON-ACCEPTANCE) of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in non-acceptance of emotional responses across the trial. The DERS was administered two times per week, and the NON-ACCEPTANCE subscale comprised 6 items with a potential score range of 6 to 30 with higher scores representing greater difficulties in acceptance of emotional response. Each time-point represents change from baseline NON-ACCEPTANCE. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties regarding non-acceptance of emotional responses compared with baseline.
Time Frame: 12-Week
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -6.4 (5.7) | -0.88 (6.6)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.08, Mixed Models Analysis

13. Secondary Outcome: Emotion Regulation (Total Score)
Description: We used the Total score of the Difficulties in Emotion Regulation Scale (DERS) to assess changes in overall emotion regulation across the trial. The DERS was administered two times per week, and comprised 41 items with a potential score range of 41 to 164 with higher scores representing greater difficulties in emotion regulation. Each time-point represents change from baseline emotion regulation difficulties. The calculation here represents mean change from baseline values across the 12 weeks, where minus values represent less difficulties regarding emotion regulation compared with baseline.
Time Frame: 12-weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
Number analyzed (Participants) | 8 | 7
scores on a scale | -19.8 (17.3) | -4.5 (21.3)
Statistical Analysis 1: Comparison: Guanfacine XR 3mgs/Daily vs Placebo (for Guanfacine); Test type: Superiority; p = 0.2, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 12-weeks
Arm/Group | Guanfacine XR 3mgs/Daily | Placebo (for Guanfacine)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7
Other Adverse Events (participants affected / at risk) | 2/8 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine XR 3mgs/Daily (N=8) | Placebo (for Guanfacine) (N=7)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) — participant admitted to ED and diagnosed with ovarian cysts
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine XR 3mgs/Daily (N=8) | Placebo (for Guanfacine) (N=7)
Headaches (General disorders) | 2 (2) | 1 (1)
Dry Mouth (General disorders) | 1 (1) | 1 (1)
Upset Stomach (General disorders) | 2 (2) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0)
Shakiness (General disorders) | 0 (0) | 1 (1)
Weight Gain (General disorders) | 1 (1) | 0 (0)
Appetite Loss (General disorders) | 1 (1) | 0 (0)
Nightmares (General disorders) | 1 (1) | 0 (0)
Enuresis (General disorders) | 1 (1) | 0 (0)
Itchiness (General disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Delay in study commencement and staff losses leading to small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT03137082/Prot_SAP_000.pdf